CLINICAL TRIAL: NCT01788462
Title: Egrifta Replacement and Sleep Disordered Breathing
Status: Withdrawn | Type: Observational
Why Stopped: Lack of funding.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Philip L. Smith ll MD, Professor of Medicine, Johns Hopkins University
Other Study IDs: NA_00074675
Record Dates: First submitted 2013-02-01; First posted 2013-02-11 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Lipodystrophy
Keywords: Tesamorelin; Egrifta; HIV; Lipodystrophy; Sleep Apnea
MeSH Terms: conditions — Lipodystrophy; Sleep Apnea Syndromes | interventions — tesamorelin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV and Lipodystrophy: The study population will consist of HIV patients with lipodystrophy who receive Tesamorelin (Egrifta).
  Interventions: Drug: Tesamorelin (Egrifta)

INTERVENTIONS:
Drug: Tesamorelin (Egrifta) — We will observe the effects of Tesamorelin on patients with HIV and lipodystrophy.
  Other Names: Egrifta TM

SUMMARY:
Sleep-disordered breathing is characterized primarily by partial or total upper airway obstruction during sleep. The most common form of sleep-disordered breathing is obstructive sleep apnea (OSA) due to recurrent collapse of the upper airway with the onset of sleep state. The major risk factors associated with the development of sleep apnea are obesity and male sex. The investigators have also found a high prevalence of OSA in HIV infected men and women, particularly among those with central lipohypertrophy, which is a common finding in HIV-infected persons receiving antiretroviral therapy. Currently, our overall hypothesis is that visceral adiposity, as seen in HIV-infected persons with central lipohypertrophy, alters both mechanical properties and compensatory neuromuscular responses leading to upper airway obstruction. Based on our most recent findings in the non-HIV population, the investigators demonstrate that obesity is associated with elevations in the upper airway load (passive Pcrit) that are counterbalanced by compensatory upper airway neural responses. Moreover, the investigators have found that female sex, peripheral adiposity, and younger age are associated with increased compensatory neuromuscular responses, while male sex, central adiposity, and older age are associated with blunted compensatory responses. The loss of the compensatory neuromuscular responses leads to obstructive sleep apnea. Among HIV-infected patients with central lipohypertrophy, tesamorelin (Egrifta), a growth hormone releasing hormone (GHRH) analogue, is approved for the reduction of visceral adipose tissue. The investigators hypothesize that tesamorelin therapy will reverse both the mechanical and neurocompensatory alterations associated with increased central obesity. In this project the investigators will determine whether tesamorelin affects sleep apnea severity and compensatory neuromuscular responses of the upper airway on sleep and breathing in men and women with HIV infection. The proposed studies are designed to elucidate the pathophysiologic basis for the development of obstructive sleep apnea in this population. The studies also provide insights into the neurohumoral regulation of upper airway function, and potentially new approaches to the treatment for sleep-disordered breathing.

ELIGIBILITY:
Inclusion Criteria:

1. Consenting adult with documented HIV-infection, ages 18 - 75 years old
2. Central lipohypertrophy as determined by a clinician
3. Not currently on Egrifta (tesamorelin) therapy.

Exclusion Criteria:

1. Unstable cardiovascular disease (decompensated CHF, myocardial infarction in past 3 months, revascularization procedure in past 3 months, and unstable arrhythmias);
2. Uncontrolled hypertension (BP > 190/110);
3. Presence of cor pulmonale
4. History of end stage renal disease (on dialysis);
5. History of end stage liver disease ( e.g. jaundice, ascites, history of recurrent gastrointestinal bleeding, transjugular intrahepatic portosystemic shunt (TIPS) ;
6. Bleeding disorders or coumadin use;
7. Tracheostomy
8. Active malignancy
9. Pregnancy and/or nursing mother -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women with HIV infection and central lipohypertrophy about to start tesamorelin therapy will be recruited from the Endocrinology Clinic at the Johns Hopkins Outpatient Center. Physicians and members of the clinical staff will identify eligible men and briefly introduce the study to them. Patients will be offered a phone number for the Johns Hopkins Sleep Disorders Center to call if they are interested in learning more about the research study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Sleep Apnea Severity | Subjects will be evaluated prior to initiating tesamorelin therapy (baseline)
  Sleep apnea severity (AHI), change in sleep apnea severity (∆ AHI), and compensatory neuromuscular responses (AT/DBT, ∆ AT/DBT) will be the primary outcome variables.
Changes in Sleep Apnea Severity | Subjects will be evaluated at three months
  Sleep apnea severity (AHI), change in sleep apnea severity (∆ AHI), and compensatory neuromuscular responses (AT/DBT, ∆ AT/DBT) will be the primary outcome variables.
Changes in Sleep Apnea Severity | Subjects will be evaluated at six months
  Sleep apnea severity (AHI), change in sleep apnea severity (∆ AHI), and compensatory neuromuscular responses (AT/DBT, ∆ AT/DBT) will be the primary outcome variables.
Changes in Sleep Apnea Severity | Subjects will be evaluated at one year
  Sleep apnea severity (AHI), change in sleep apnea severity (∆ AHI), and compensatory neuromuscular responses (AT/DBT, ∆ AT/DBT) will be the primary outcome variables.

SECONDARY OUTCOMES:
Changes in Body Composition | baseline
  Secondary outcomes will include the percent change in anthropometric and body composition parameters as reflected by Dual-Energy Xray Absorbtiometry measurements.
Changes in Body Composition | 12 months
  Secondary outcomes will include the percent change in anthropometric and body composition parameters as reflected by Dual-Energy Xray Absorbtiometry measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Philip L Smith, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Sleep Disorders Center, Baltimore, Maryland, United States